CLINICAL TRIAL: NCT00045513
Title: Phase I/II Study Of UCN-01 In Combination With Fludarabine In Patients With Relapsed Or Refractory Chronic Lymphocytic Leukemia Or Small Lymphocytic Lymphoma
Brief Title: Combination Chemotherapy in Treating Patients With Chronic Lymphocytic Leukemia or Lymphocytic Lymphoma
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Purpose: Treatment
Other Study IDs: PMH-PHL-006; CDR0000256600 (Registry Identifier: PDQ (Physician Data Query)); NCI-5538
Record Dates: First submitted 2002-09-06; First posted 2003-01-27 (Estimated); Last update posted 2015-07-23 (Estimated); Status verified 2015-07

CONDITIONS: Leukemia; Lymphoma
Keywords: refractory chronic lymphocytic leukemia; recurrent small lymphocytic lymphoma
MeSH Terms: conditions — Leukemia; Lymphoma; Leukemia, Lymphocytic, Chronic, B-Cell | interventions — 7-hydroxystaurosporine; fludarabine phosphate

INTERVENTIONS:
Drug: 7-hydroxystaurosporine
Drug: fludarabine phosphate

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop cancer cells from dividing so they stop growing or die. Combining more than one drug may kill more cancer cells.

PURPOSE: Phase I/II trial to study the effectiveness of combining UCN-01 with fludarabine in treating patients who have relapsed or refractory chronic lymphocytic leukemia or lymphocytic lymphoma.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the overall response rate in patients with relapsed or refractory chronic lymphocytic leukemia (CLL) or small lymphocytic lymphoma treated with UCN-01 and fludarabine.
* Assess the molecular changes in CLL cells in peripheral blood in patients treated with this regimen.
* Determine the progression-free and overall survival of patients treated with this regimen.
* Determine the toxicity of this regimen in these patients.

OUTLINE: This is a multicenter, dose-escalation study of UCN-01.

Patients receive UCN-01 IV over 3 hours on day 1 and fludarabine IV over 30-60 minutes on days 1-5. Treatment repeats every 4 weeks for up to 6 courses in the absence of disease progression or unacceptable toxicity.

Cohorts of 3-6 patients receive escalating doses of UCN-01 until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which at least 2 of 3 or 2 of 6 patients experience dose-limiting toxicity. Once the MTD is determined, 18-46 additional patients receive UCN-01 and fludarabine as above at the recommended phase II dose.

PROJECTED ACCRUAL: A total of 12 patients will be accrued for the phase I portion of this study within 6 months. A total of 18-46 patients will be accrued for the phase II portion of this study within 9-23 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically confirmed chronic lymphocytic leukemia (CLL) or B-cell small lymphocytic lymphoma (SLL)

  * CLL is defined as:

    * Persistent lymphocytosis greater than 5,000/mm^3
    * CD19/CD5/CD23 positive
    * Kappa or lambda light chain restriction
* Refractory to or disease progression after 1 or 2 prior treatment regimens

  * Retreatment with oral chlorambucil is allowed and considered a second regimen

    * At least one of the chlorambucil treatments must be for 3 months or longer
  * At least 4 courses of cyclophosphamide, vincristine, and prednisone with or without doxorubicin allowed
  * Patients may have received prior fludarabine as first- or second-line therapy if there is evidence of at least partial response and time to progression after initial fludarabine therapy was at least 12 months
* No CNS involvement by lymphoma

PATIENT CHARACTERISTICS:

Age

* 18 and over

Performance status

* ECOG 0-2 OR
* Karnofsky 60-100%

Life expectancy

* More than 3 months

Hematopoietic

* See Disease Characteristics
* Absolute neutrophil count at least 1,000/mm^3
* Platelet count at least 100,000/mm^3
* No autoimmune hemolytic anemia or thrombocytopenia secondary to CLL or SLL requiring ongoing therapy with prednisone or other immunosuppressive agents

Hepatic

* Bilirubin normal
* AST and ALT no greater than 2.5 times upper limit of normal

Renal

* Creatinine normal OR
* Creatinine clearance at least 60 mL/min

Cardiovascular

* No symptomatic congestive heart failure
* No unstable angina pectoris
* No cardiac arrhythmia

Pulmonary

* DLCO greater than 60% predicted
* FEV_1 greater than 70% predicted
* No significant underlying pulmonary disease

Other

* No other malignancy within the past 5 years except adequately treated basal cell skin cancer or carcinoma in situ of the cervix
* No insulin-dependent diabetes mellitus
* No other uncontrolled concurrent illness
* No ongoing or active infection
* No pre-existing peripheral neuropathy grade 2 or greater
* No psychiatric illness or social situation that would preclude study compliance
* No prior allergic reactions to compounds of similar chemical or biological composition to UCN-01 or other agents in this study
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY:

Biologic therapy

* Not specified

Chemotherapy

* See Disease Characteristics
* At least 4 weeks since prior chemotherapy and recovered

Endocrine therapy

* See Hematopoietic

Radiotherapy

* No prior mediastinal radiation
* At least 4 weeks since prior radiotherapy and recovered

Surgery

* Not specified

Other

* No other concurrent investigational agents
* No concurrent combination antiretroviral therapy for HIV-positive patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2002-06; Primary Completion 2003-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael R. Crump, MD, FRCPC, Study Chair — Princess Margaret Hospital, Canada
Locations (3):
- Canada (3):
  - McMaster Children's Hospital at Hamilton Health Sciences, Hamilton, Ontario
  - London Health Sciences Centre, London, Ontario
  - Princess Margaret Hospital at University Health Network, Toronto, Ontario